CLINICAL TRIAL: NCT03360383
Title: Effect and Essentiality of Vertebroplasty Surgery in Acute Vertebral Compression Fractures: a Multiple Center Randomized Controlled Trial
Brief Title: Effect and Essentiality of Vertebroplasty Surgery in Acute Vertebral Compression Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Liu Haiying, Director department of spinal surgery, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AVCF1
Record Dates: First submitted 2017-11-25; First posted 2017-12-04 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-12

CONDITIONS: Spinal Fractures
Keywords: Spinal Fractures/surgery; Vertebroplasty; Quality-Adjusted Life Years
MeSH Terms: conditions — Spinal Fractures | interventions — Conservative Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- grade 1 (Experimental): percutaneous vertebroplasty
  Interventions: Procedure: percutaneous vertebroplasty
- grade 2 (Active Comparator): conservative treatment
  Interventions: Procedure: conservative treatment

INTERVENTIONS:
Procedure: percutaneous vertebroplasty — Undertake Percutaneous vertebroplasty with polymethylmetacrylate bone cement.
  Arms: grade 1
Procedure: conservative treatment — complete on bed with prevention of complications
  Arms: grade 2

SUMMARY:
Percutaneous vertebroplasty is now a common procedures of patients with acute osteoporotic vertebral compression fractures in medical units all over China, but the efficacy and essentiality of the surgery remain uncertain and is the subject of this study. This is a multiple center open-label randomised trial. Patients were randomly allocated to percutaneous vertebroplasty or conservative treatment. Because of the procedure , neither patients nor investigators were blinded. The primary outcome was pain relief at 1 month and 1 year.

DETAILED DESCRIPTION:
This study will use a randomised controlled trial to access the efficacy and essentiality of the surgery for vertebral compression fractures. Patients aged 50 years or older, had vertebral compression fractures on spine radiograph (minimum 15% height loss) will be invited to take part. Patients will be randomised into 2 arms with average amount. The participants in the intervention arm will have percutaneous vertebroplasty ; those randomised to the control arm will receive current standard conservative treatment methods.

Patients were clinically assessed at baseline (the day of surgery or treatment), and at 1 day, 1 week, 1 month, 3 months, 6 months, and 1 year afterwards. The primary outcome will be the pain release , categorised according to WHO classification.

ELIGIBILITY:
Inclusion Criteria:

* vertebral compression fracture on spine radiograph (minimum 15% height loss)
* level of fracture at Th5 or lower; back pain for 6 weeks or less
* focal tenderness at fracture level on physical examination
* bone oedema of vertebral fracture on MRI
* decreased bone density (T scores ≤-1)

Exclusion Criteria:

* severe cardiopulmonary comorbidity
* suspected underlying malignant disease
* radicular syndrome
* spinal-cord compression syndrome
* contraindication for radiography exam

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2018-02-01 (Estimated); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
change of pain relief | 1 day, 1 week, 1 month, 3 months, 6 months, and 1 year
  World Health Organization pain classification

SECONDARY OUTCOMES:
quality of life | 1 day, 1 week, 1 month, 3 months, 6 months, and 1 year
  Quality of Life Questionnaire of the European Foundation for Osteoporosis (QUALEFFO)

CONTACTS AND LOCATIONS:
Overall Officials: haiying liu, Study Director — PekingUPH department of spinal surgery

IPD SHARING:
Plan to Share IPD: No